CLINICAL TRIAL: NCT02483533
Title: A Double-Blind Extension Study to Evaluate the Post-Treatment Safety and Duration of Clinical Effect of LIPO-202 in Subjects Who Completed Either the LIPO-202-CL-18 or LIPO-202-CL-19 Study
Brief Title: Extension Study to Evaluate the Post-Treatment Safety and Duration of Clinical Effect of LIPO-202
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Evofem Inc. (Industry)
Collaborators: Neothetics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: LIPO-202-CL-23
Record Dates: First submitted 2015-06-17; First posted 2015-06-29 (Estimated); Results first posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-11

CONDITIONS: Central Abdominal Bulging

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental: LIPO-202 (Experimental): Subjects received either LIPO-202 or Placebo for LIPO-202 in the parent study (LIPO-202-CL-18 or LIPO-202-CL-19). Subjects will not receive any additional treatment in this follow-on study.
  Interventions: Drug: LIPO-202
- Placebo Comparator: Placebo (Placebo Comparator): Subjects received either LIPO-202 or Placebo for LIPO-202 in the parent study (LIPO-202-CL-18 or LIPO-202-CL-19). Subjects will not receive any additional treatment in this follow-on study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LIPO-202
  Arms: Experimental: LIPO-202
Drug: Placebo
  Other Names: Placebo for LIPO-202
  Arms: Placebo Comparator: Placebo

SUMMARY:
LIPO-202-CL-23 is a follow-on study to evaluate the post-treatment safety and duration of clinical effect of LIPO-202 in subjects that completed either the LIPO-202-CL-18 (NCT02397499) or LIPO-202-CL-19 (NCT02398188). No risks related to treatment are anticipated as subjects will not receive additional treatment with LIPO-202 or Placebo for LIPO-202 in this follow-on study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female subjects who completed Study LIPO-202-CL-18 or LIPO-202-CL-19
* Capable of providing written consent
* Willing to comply with the study procedures and schedule

Exclusion Criteria:

* Female subjects who are pregnant or are not using adequate birth control methods
* Plan on starting a weight loss or exercise program during the study
* Plan to enroll in another investigational drug or device study
* Unlikely or unable to adhere to the study visit schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12-23 (Actual); Study Completion 2016-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Feldman, Study Director — Neothetics, Inc

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: LIPO-202: Subjects received either LIPO-202 or Placebo for LIPO-202 in the parent study (LIPO-202-CL-18 or LIPO-202-CL-19). Subjects will not receive any additional treatment in this follow-on study.
  LIPO-202
- Placebo Comparator: Placebo: Subjects received either LIPO-202 or Placebo for LIPO-202 in the parent study (LIPO-202-CL-18 or LIPO-202-CL-19). Subjects will not receive any additional treatment in this follow-on study.
  Placebo
Period: Overall Study
Arm/Group | Experimental: LIPO-202 | Placebo Comparator: Placebo
Started (Lack of efficacy - not completed) | 50 | 50
Completed (Lack of efficacy - not completed) | 0 | 0
Not Completed | 50 | 50
Not completed — Lack of Efficacy | 50 | 50

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: LIPO-202 | Placebo Comparator: Placebo | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of the Post-treatment Duration of Clinical Effect of LIPO-202. Photonumeric Score and Global Abdominal Perception Score.
Description: Measured by change in clinician reported photonumeric score and change in patient reported global abdominal perception score. Patient-rated changes in amount of bulging or flatness of their belly using the 5-point scale provided as pictures where zero is flat and five is big bulge.
Time Frame: 1 Year
Population: Lack of efficacy - not completed. Study was conducted by Neothetics Inc. and during a company merger with Evofem, no study data was provided. All efforts to locate this data have been exhausted, there is no longer access to this data to be reported.
Arm/Group | Experimental: LIPO-202 | Placebo Comparator: Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Evaluation of a 12-month Post-treatment, Non-interventional, Observational Period to Evaluate the Safety and Duration of Clinical Effects of LIPO-202.
Description: Subjects who report an improvement of a least 1-point (grade) on the patient global abdominal perception scale and the photonumeric scale.
Time Frame: 1 Year
Population: as for outcome 1
Arm/Group | Experimental: LIPO-202 | Placebo Comparator: Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Experimental: LIPO-202 | Placebo Comparator: Placebo
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No